CLINICAL TRIAL: NCT05826769
Title: To Assess the Efficacy of Early Administration of Energy Enriched and Protein Enriched Formula in Post Cardiac Repair Infants: a Randomized Controlled Trial, Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-34
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease in Children; Post-cardiac Surgery; Malnutrition, Infant
Keywords: Energy Protein, Enriched; Enteral Nutrition; Cardiac Repair
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: * Patients are randomized before surgery in blocks of 2 using a computer-generated randomization list into intervention and control groups
  * This will be An open, 2-arm,randomized controlled trial
Masking Description: According to national regulations, distribution of infant formula inside the hospital without a proper label is not allowed; therefore, subjects can not be blinded in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy- Protein Enriched Nutritional Formula (Experimental): Liquid, ready-to-use Energy-Protein nutrition formula with energy density of 1 kCal/mL (EP formula)
  Interventions: Dietary Supplement: Energy- Protein Enriched Nutritional Formula
- Standard Nutritional Formula (No Intervention): Polymeric formula stage-1 and stage-2 for infants aged 0-6 months and 6-12 months accordingly, providing 0.67 kCal/mL (S-1/S-2 formula)

INTERVENTIONS:
Dietary Supplement: Energy- Protein Enriched Nutritional Formula — EN volume will start at 1 mL/kg/h and then increase by 1 mL/kg every 6 hours if tolerated, until reaching 130 mL/kg/d.
  Other Names: High Calorie High Protein Nutritional Formula
  Arms: Energy- Protein Enriched Nutritional Formula

SUMMARY:
Congenital heart disease (CHD) is a public health problem, A substantial percentage of infants and toddlers with CHD undergo cardiopulmonary bypass surgery. Undernutrition affects up to 90% of these patients, and it's contributed to worse surgical and neurological outcomes. Infants with CHD are typically delivered at full term with a normal birth weight. However, as time passes, their development may become stunted. There are no negotiated guidelines for nutritional monitoring and intervention in this age bracket of infants. Through the use of Energy Enriched and Protein Enriched nutrition formula during the postoperative phase, this has shown to be well tolerated and support in delivering higher nutrition intakes within the first days after surgery. The objective of this research is to assess the long term outcome of patients who have had energy- and protein-rich nutrition formulas post cardiac surgery. An open, 2-arm, randomized controlled trials will be conducted to assess the efficacy of early administration of energy enriched and protein enriched formula in post cardiac repair infants. The expected primary outcome is that intervention group will have good tolerance to feeding and the secondary outcome is the significant weight gain rate (weight velocity) in comparing to control groups

DETAILED DESCRIPTION:
Due to a high incidence of 9/1000 live births, congenital heart disease (CHD) is a public health problem, A substantial percentage of infants and toddlers with CHD undergo cardiopulmonary bypass surgery. Undernutrition affects up to 90% of these patients, and it's contributed to worse surgical and neurological outcomes. Infants with CHD are typically delivered at full term with a normal birth weight. However, as time passes, their development may become stunted. There are no negotiated guidelines for nutritional monitoring and intervention in this age bracket of infants. Through the use of Energy Enriched and Protein Enriched nutrition formula during the postoperative phase, this has shown to be well tolerated and support in delivering higher nutrition intakes within the first days after surgery. Numerous clinical trials have been conducted (Zhang H et al., 2018; Scheeffer. et al., 2019) and were designed to explore the effects of early introduction of Energy Enriched and Protein Enriched formula (EP) to infants with CHD. The research found that feeding EP is correlated with improved weight gain and nutritional status, and also a decrease in Hospital Length Of Stay (HLOS) as well as antibiotic use, but this also causes increased feeding discomfort. The signs of feeding discomfort, on the other hand, were improved by medication and had little effect on feeding progress.

The objective of this research is to assess the long term outcome of patients who have had energy- and protein-rich nutrition formulas post cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. infants born at term, age between 4 weeks and 12 months
2. post congenital heart surgery (RACHS score 2)

Exclusion Criteria:

1. syndromic patients
2. if patient is on parenteral nutrition (PN)
3. premature
4. combined inherited metabolic or chromosomal diseases
5. liver and kidney dysfunction before enrollment (index >2 times the upper limit of normal)
6. upper GI activity, vomiting, diarrhea, bloating, and other symptoms before enrollment
7. breastfeeding patients.
8. cow's milk allergy

Ages: 4 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
after admission in ICU, will measure the Tolerability | 5 days
  Gastric tolerance

SECONDARY OUTCOMES:
Weight gain rate | 90 days
  Weight velocity

CONTACTS AND LOCATIONS:
Locations (1):
- KFSHRC, Jeddah, Outside North America, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided